CLINICAL TRIAL: NCT00133926
Title: Prevention of Pre-Term Birth by Treatment of Periodontal Disease During Pregnancy - The Smile Study
Brief Title: Prevention of Pre-Term Birth by Treatment of Periodontal Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Memorial Hospital (Other)
Collaborators: The University of Western Australia (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 353577; NHMRC Australia 353577
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Periodontal Diseases; Premature Birth; Pre-Eclampsia
Keywords: Periodontal disease; Pregnancy; Pre-term birth; Fetal growth; Pre-eclampsia; Infant, Low Birth Weight
MeSH Terms: conditions — Periodontal Diseases; Premature Birth; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Treatment of periodontal disease

SUMMARY:
The aim of the study is to investigate, in an Australian population of pregnant women, whether the treatment of periodontal disease during pregnancy prevents pre-term birth and other complications of pregnancy. Dental screening and periodontal treatment protocols have been based on standard techniques employed by hygienists that can be readily applied to the general obstetric population.

DETAILED DESCRIPTION:
HYPOTHESES

Primary Hypothesis:

That treatment of periodontal disease during pregnancy reduces the rate of pre-term birth from 12% to 7%.

Secondary Hypothesis:

That treatment of periodontal disease during pregnancy reduces the rate of:

* Fetal growth restriction.
* Complications of pre-term birth including respiratory distress syndrome.
* Periodontal disease measured at 36 weeks gestation.

Research Plan Synopsis:

A randomized controlled trial is being conducted with recruitment of women from the antenatal clinics of Perth's major obstetric centres and associated private practices. The sample is being enriched by inviting women with a history of poor oral health or pre-term birth. 5400 eligible women will undergo a hygienist-based screening study at 12-20 weeks gestation. 1094 women who meet the criteria for periodontal disease determined from our recent pilot study will be allocated at random to the treatment or control groups. Those in the treatment group will receive three one-hour hygienist-based periodontal treatment sessions commencing at 20 weeks gestation, followed by re-examination at 26 weeks. Re-treatment will be offered to the 5% of cases in which treatment has been ineffective, and ongoing maintenance to the remainder. Women allocated to the control group will be offered similar treatment after completion of the pregnancy.

RESEARCH PLAN

Study Design:

Multi-centered single-blinded randomized controlled trial conducted within the metropolitan area of Perth, Western Australia. The obstetric and newborn health care providers are blinded to the periodontal treatment allocation.

Inclusion Criteria:

Women with single pregnancies at 12 to 20 weeks gestation with periodontal disease defined as periodontal pocketing at a threshold of 4mm or more at 10% or more of sites and who agree to receive periodontal treatment are eligible. The definition of periodontal disease is based on the published literature and our pilot study designed to determine the prevalence in our local obstetric population. Periodontal pocketing is used to define the presence of periodontal disease rather than clinical loss of attachment because it better represents the microbial challenge and is the most frequently employed criterion. In our pilot study, 15% of our general unselected population met this criterion.

Exclusion Criteria:

Women are ineligible if they are: unable to attend for periodontal treatment; less than 16 years of age; present for antenatal care after 20 weeks gestation; are unable to understand the implications of participation in the trial; have a fetus with a known abnormality that would predispose the pregnancy to pre-term birth such as those that may cause polyhydramnios; have a multiple pregnancy; have cardiac disease that would require antibiotic therapy for dental treatment; are currently receiving periodontal treatment; or have fewer than 20 teeth.

Trial Entry:

All women planning to attend the antenatal clinics at King Edward Memorial Hospital (KEMH) in Perth, Western Australia are provided with written information about the trial with their appointment letter. Those attending other public antenatal clinics and a proportion of private practices also receive the information and invitation. Women who do not have exclusion criteria are invited by a research midwife to provide written informed consent to undergo a periodontal examination. After the examination those women who meet the criteria for periodontal disease are invited by a member of the research team to participate in the trial and to provide written informed consent to have treatment. A questionnaire is administered to obtain data on demographic and medical factors that may influence oral health and details of past and present dental care. Women who are found to not have periodontal disease are asked to provide consent for their obstetric outcomes to be retrieved from the state-wide computerized data collection system that encompasses all births in Western Australia.

Randomisation:

Each woman is allocated to the treatment or control group by the sealed-envelope technique, prepared in blocks of 20. Recruitment is stratified by history of pre-term birth, nulliparity and smoking practice. Women who smoke in either arm of the study are provided with written material encouraging them to cease smoking.

Management of the Treatment Group:

Women allocated to the treatment group are given appointments to attend the Oral Health Centre of Western Australia (OHCWA).

Management of the Control Group:

Women allocated to the control group are provided with the findings of their periodontal examination to take to their dentist and written information on oral health care. Each woman is also invited to receive free dental care at OHCWA commencing 6 weeks after delivery and continuing for 16 weeks, as described below.

Dental Examination:

The simple screening dental examination is a modified WHO CPITN (Gjermo,1998) conducted in a well-equipped dental room within the antenatal clinic at KEMH. This examination takes approximately 20 minutes and is conducted by a study hygienist under supervision by the study periodontists. If periodontitis is detected the woman is invited to participate in the trial as described previously.

Periodontal Treatment:

Treatment Group:

All periodontal treatment is conducted in the Oral Health Centre of Western Australia (OHCWA), located 2 km from KEMH. A full periodontal examination is first performed using a constant force automated Florida probe (Florida Probe Corporation, Gainesville, Florida, USA) which provides precise measurements of pocket depth to 0.2mm, and stores data directly into a computer. This measurement system has been used in our pilot study and two separate probes and computer systems are available for this trial. Further periodontal parameters are recorded, including clinical attachment loss, full mouth bleeding after probing, and modified O'Leary Plaque Index. Treatment explanation is then provided by the hygienist and consent confirmed. The treatment plan for each woman is determined in consultation with a study periodontist and is conducted over 3 visits each of one hour duration. These treatments consist of non-surgical debridement of the sub- and supra-gingival plaque, removal of local predisposing factors such as calculus, and adjustment of overhanging restorations. Comprehensive oral hygiene instruction and motivation is provided at each visit as required. This oral hygiene advice recommends tooth brushing and flossing after every meal and rinsing with 0.12% non-alcohol based chlorhexidine mouth wash. These treatments are provided on 3 occasions at weekly intervals commencing at 20 weeks gestation.

Local anaesthesia is employed as required (1% lignocaine with 1:80,000 adrenalin up to a maximum dose of 10mls).

Four weeks after the final treatment, at approximately 28 weeks gestation, a further visit is made to re-evaluate periodontal status using clinical examination and the Florida probe. This examination provides a quantifiable assessment of the success of treatment. Those women in whom treatment has been unsuccessful are offered a further 3-visit treatment plan and we estimate this will be required in 5-10% of the sample. A further two visits, each of 45 minutes duration is scheduled for 32 and 36 weeks gestation, at which times periodontal supportive care and oral hygiene instruction and motivation are carried out as required. Periodontal parameters at these visits are recorded.

Full infection control barrier techniques are employed and are stringent. Procedures include gowns, disposable gloves and masks, eye protection for examiner and patient, and barrier methods to avoid contamination.

Systemic antibiotic treatment is not employed except in cases in which there is evidence of multiple periodontal abscesses, impaired immune response or poorly controlled diabetes. In such cases treatment involves oral metronidazole and amoxycillin in standard doses for 5 days commencing with the treatment. In the pilot study we observed no cases meeting these criteria.

Control Group:

Women allocated to the control group are offered periodontal care after birth commencing 6 weeks after delivery. This care involves the same initial assessment and 3-visit treatment protocol as for women in the treatment group. A further full periodontal examination is conducted 4 weeks later.

After completion of their involvement in the study, women in both groups will be offered ongoing maintenance care at OCHWA and this care will be free of charge if they hold a health care card.

Women Who Deliver Pre-Term:

Those women who deliver pre-term will be offered a further screening examination at OHCWA and treatment as for the control group. Information in this regard will be provided at the time of recruitment.

Obstetric Management:

The obstetric and midwifery health care providers are unaware of the treatment allocation of each woman in the study. Care is provided according to the standard protocols employed within each hospital.

Sample Size:

The sample is enriched by advertising in the general media and in our peripheral public hospitals for women with poor oral health or a history of pre-term birth to attend KEMH for a single visit between 12 and 20 weeks gestation for periodontal examination.

A sample size of 540 women in each arm provides power to detect a reduction in the rate of pre-term birth from 12% to 7% with power of 90% and an alpha level of 5%. Our pilot study of 272 women revealed a rate of periodontal disease of 15% in unselected women. With enrichment by advertising for women at higher risk, we estimate the rate of periodontal disease will be 20%. Thus, for a total study size of 1080 women, 5400 need to be screened, which is rate of 45 each week in a 48 week working year. This sample size estimate allows two interim analyses.

Statistical Considerations:

A data monitoring committee will be formed and will include an independent statistician who will conduct the interim analysis. The committee will cease the trial if pre-determined rates of benefit or harm are achieved. Analyses will be conducted on an intention-to-treat basis using tests of proportions and logistic regression that allow for multiple adjustment for covariates. Secondary analyses will be conducted of dose-response of treatment and appropriate comparisons made with women who received periodontal examinations but did not meet eligibility criteria. All hypothesis testing will be two sided and significance will be at the 5% level.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, with single pregnancies, between 12 and 20 weeks gestation
* Periodontal disease defined as periodontal pocketing at a threshold of 4mm or more at 10% or more of sites
* Agree to receive periodontal treatment

Exclusion Criteria:

* Unable to attend for treatment
* Less than 16 years of age
* Have a fetus with an abnormality that predisposes the pregnancy to pre-term birth
* Multiple pregnancy
* Cardiac disease that would require antibiotic therapy
* Have fewer than 20 teeth
* Present for antenatal care after 20 weeks gestation
* Unable to understand the implications of participation in the trial
* Currently receiving periodontal treatment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1094
Dates: Start 2005-03; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Rate of pre-term birth

SECONDARY OUTCOMES:
Rate of fetal growth restriction
Rate of pre-eclampsia
Rate of complications of pre-term birth

CONTACTS AND LOCATIONS:
Overall Officials: John P Newnham, MD, FRANZCOG, Principal Investigator — The University of Western Australia
Locations (1):
- King Edward Memorial Hospital, Bagot Rd, Subiaco, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Newnham JP, Newnham IA, Ball CM, Wright M, Pennell CE, Swain J, Doherty DA. Treatment of periodontal disease during pregnancy: a randomized controlled trial. Obstet Gynecol. 2009 Dec;114(6):1239-1248. doi: 10.1097/AOG.0b013e3181c15b40. PMID 19935025